CLINICAL TRIAL: NCT03452865
Title: Proton Pump Inhibitors (PPI) as a New Strategy for Therapy in Sepsis: Clinical Trial to Reduce Severity of Organ Failure and in Vitro Experiments to Search Specific Hallmarks in Monocytes From Septic Patients and to Characterize the Mechanism of Action of PPI
Brief Title: Esomeprazole to Reduce Organ Failure in Sepsis
Acronym: PPI-SEPSIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPI-SEPSIS; 2018-000488-98 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Septic Shock
Keywords: proton pump inhibitor; esomeprazole; sepsis; septic shock; organ failure; SOFA; mortality
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esomeprazole (Experimental): Patients randomized to Esomeprazole Group will receive a bolus of 160 mg of esomeprazole (diluted in 100 ml of 0.9% sodium chloride for intravenous use and administered over 60 minutes) and an intravenous infusion of 12 mg/hr (diluted in 0.9% sodium chloride at a concentration of 8 mg/ml will be injected at a rate of 1.5 ml/hr) for 72 hours .
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator): Patients randomized to Placebo Group will receive a bolus of 100 ml of 0.9% sodium chloride for intravenous use administered over 60 minutes with no active principle and an intravenous infusion of 0.9% sodium chloride at a rate of 1.5 ml/hr with no active principle for 72 hours .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 160 mg of esomeprazole will be diluted in 100 ml of 0.9% sodium chloride for intravenous use for bolus.
  For continuous intravenous infusion, 40 mg of esomeprazole will be reconstituted by adding 5 ml of 0.9% sodium chloride for intravenous use at a concentration of 8 mg/ml.
  Arms: Esomeprazole
Drug: Placebo — 0.9% sodium chloride (same ml of the study drug)
  Arms: Placebo

SUMMARY:
Sepsis is a severe disease with a high mortality rate and lack of efficacious therapies. Proton pump inhibitors (PPI) are drugs widely used to inhibit acid secretion by gastric cells and with a high safety profile. Carta and Rubartelli (IRCCS San Martino - Genova) have recently reported that PPI, such as esomeprazole, inhibit TNF-alfa and IL-1ß secretion. Moreover, they showed that a single administration of PPI protects mice from endotoxic shock with no adverse effects. PPI-SEPSIS is a randomized, double blind, controlled against placebo clinical trial to test if high-doses esomeprazole in septic patients reduces the severity of organs failure.

In parallel, the investigators will evaluate ex vivo in monocytes from septic patients: redox state and response to inflammatory stimuli; ATP release; metabolic changes and pH; cytokine production; the effects of PPI on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Admitted to intensive care unit or emergency department
* Sepsis or septic shock
* Able to express informed consent. For unconscious patients, current laws will be applied as requested by Ethical Committee.

Exclusion Criteria

* Able to express informed consent and deny it
* Known allergy or intolerance to study drug
* Little chance of survival, as defined by a SAPS II score more than 65 point
* Concomitant acquired immunodeficiency syndrome
* On immunosuppressant or long-term corticosteroid therapy
* Receiving lifesaving drugs known to have a strong interference with esomeprazole
* Sepsis or septic shock since over 36 hours
* Severe hepatic dysfunction
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
SOFA score reduction | Days 1-28
  SOFA (sequential organ failure assessment) score is used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems which are added up. Each score ranges from 0 to 4. SOFA score ranges from 0 (better outcome) to 24 points (worse outcome).

SECONDARY OUTCOMES:
Mortality | Day 28, 60 and 90
Antibiotic-free days | Day 28
Adjusted ICU-free days | Day 28
Single organ failure severity | Days 1-28
  Highest mean difference in each different category of SOFA score. SOFA (sequential organ failure assessment) score is used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems which are added up. Each score ranges from 0 to 4. SOFA score ranges from 0 (better outcome) to 24 points (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Monti, MD, Principal Investigator — Department of Anesthesia and Intensive Care, IRCCS San Raffaele Scientific Institute; Giovanni Landoni, MD, Study Chair — Associate Professor of Anesthesiology and Intensive Care, Vita-Salute San Raffaele University
Locations (17):
- Italy (14):
  - Policlinico Univeristario Campus Bio-Medico, Rome, Lazio
  - IRCCS San Martino Istitute, Genoa, Liguria
  - Humanitas Clinical Institute, Rozzano, Lombardy
  - IRCCS San Raffaele Scientific Institute, Milan, MI
  - A.O.U. Mater Domini, Catanzaro, Reggio Calabria
  - Azienda Ospedaliera Universitaria, Cagliari, Sardinia
  - USSL 10 Veneto, San Donà di Piave, Venezia
  - Ospedale Maggiore di Lodi, Lodi
  - Ospedale di Merano, Merano
  - Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - AOU Pisana, Pisa
  - A.O.R San Carlo, Potenza
  - Azienda Ospedaliera San Giovanni Battista Molinette di Torino, Torino
  - Ospedale Santa Maria della Misericordia, Udine
- Astana Medical University, Kazakhstan, Kazakhstan
- Russia (2):
  - Federal Clinical & Research Center for Reanimatology and Rehabilitation, Moscow
  - Negovskiy Reanimatology Research Institute, Moscow

REFERENCES:
- [Background] Mayr FB, Yende S, Angus DC. Epidemiology of severe sepsis. Virulence. 2014 Jan 1;5(1):4-11. doi: 10.4161/viru.27372. Epub 2013 Dec 11. PMID 24335434
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Ferner RE, Allison TR. Omeprazole overdose. Hum Exp Toxicol. 1993 Nov;12(6):541-2. doi: 10.1177/096032719301200614. PMID 7904473
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Background] Forrester MB. Pattern of proton pump inhibitor calls to Texas poison centers, 1998-2004. J Toxicol Environ Health A. 2007 Apr 15;70(8):705-14. doi: 10.1080/15287390601188045. PMID 17365625
- [Background] Neumann I, Letelier LM, Rada G, Claro JC, Martin J, Howden CW, Yuan Y, Leontiadis GI. Comparison of different regimens of proton pump inhibitors for acute peptic ulcer bleeding. Cochrane Database Syst Rev. 2013 Jun 12;2013(6):CD007999. doi: 10.1002/14651858.CD007999.pub2. PMID 23760821
- [Background] Orme RM, Perkins GD, McAuley DF, Liu KD, Mason AJ, Morelli A, Singer M, Ashby D, Gordon AC. An efficacy and mechanism evaluation study of Levosimendan for the Prevention of Acute oRgan Dysfunction in Sepsis (LeoPARDS): protocol for a randomized controlled trial. Trials. 2014 Jun 2;15:199. doi: 10.1186/1745-6215-15-199. PMID 24894386
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- [Background] Noritomi DT, Soriano FG, Kellum JA, Cappi SB, Biselli PJ, Liborio AB, Park M. Metabolic acidosis in patients with severe sepsis and septic shock: a longitudinal quantitative study. Crit Care Med. 2009 Oct;37(10):2733-9. doi: 10.1097/ccm.0b013e3181a59165. PMID 19885998
- [Background] Balza E, Piccioli P, Carta S, Lavieri R, Gattorno M, Semino C, Castellani P, Rubartelli A. Proton pump inhibitors protect mice from acute systemic inflammation and induce long-term cross-tolerance. Cell Death Dis. 2016 Jul 21;7(7):e2304. doi: 10.1038/cddis.2016.218. PMID 27441656
- [Background] Lavieri R, Piccioli P, Carta S, Delfino L, Castellani P, Rubartelli A. TLR costimulation causes oxidative stress with unbalance of proinflammatory and anti-inflammatory cytokine production. J Immunol. 2014 Jun 1;192(11):5373-81. doi: 10.4049/jimmunol.1303480. Epub 2014 Apr 25. PMID 24771848
- [Background] Cui LH, Li C, Wang XH, Yan ZH, He X, Gong SD. The therapeutic effect of high-dose esomeprazole on stress ulcer bleeding in trauma patients. Chin J Traumatol. 2015;18(1):41-3. doi: 10.1016/j.cjtee.2014.06.001. PMID 26169094
- [Derived] Monti G, Carta S, Kotani Y, Bruni A, Konkayeva M, Guarracino F, Yakovlev A, Cucciolini G, Shemetova M, Scapol S, Momesso E, Garofalo E, Brizzi G, Baldassarri R, Ajello S, Isirdi A, Meroi F, Baiardo Redaelli M, Boffa N, Votta CD, Borghi G, Montrucchio G, Rauch S, D'Amico F, Pace MC, Paternoster G, Vitale F, Giardina G, Labanca R, Lembo R, Marmiere M, Marzaroli M, Nakhnoukh C, Plumari V, Scandroglio AM, Scquizzato T, Sordoni S, Valsecchi D, Agro FE, Finco G, Bove T, Corradi F, Likhvantsev V, Longhini F, Konkayev A, Landoni G, Bellomo R, Zangrillo A; PPI-SEPSIS Study Group. A Multinational Randomized Trial of Mega-Dose Esomeprazole as Anti-Inflammatory Agent in Sepsis. Crit Care Med. 2025 Aug 1;53(8):e1554-e1566. doi: 10.1097/CCM.0000000000006720. Epub 2025 May 29. PMID 40439536
- [Derived] Monti G, Konkayev A, Carta S, Bradic N, Bruni A, Kotani Y, Guarracino F, Redkin I, Biondi-Zoccai G, Benedetto U, D'Ascenzo F, Garofalo E, Baiardo Redaelli M, Brizzi G, Forfori F, Borghi G, Scapol S, Momesso E, Cuffaro R, Boffa N, Rauch S, D'Amico F, Montrucchio G, Pace MC, Galbiati C, Bosso S, Savelli F, Giardina G, Silvetti S, Tripodi VF, Labanca R, Lembo R, Marmiere M, Marzaroli M, Nakhnoukh C, Valsecchi D, Finco G, Agro FE, Bove T, Corradi F, Longhini F, Landoni G, Bellomo R, Zangrillo A; Collaborators. High dose esomeprazole as an anti-inflammatory agent in sepsis: Protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Oct;133:107319. doi: 10.1016/j.cct.2023.107319. Epub 2023 Aug 23. PMID 37625587